CLINICAL TRIAL: NCT06762938
Title: The Effect of ShotBlocker on Pain and Satisfaction During Measles-Rubella-Mumps Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Veysel Can, Asst. Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: ShotBlocker
Record Dates: First submitted 2024-12-31; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ShotBlocker (Experimental)
  Interventions: Behavioral: ShotBlocker
- Control (No Intervention)

INTERVENTIONS:
Behavioral: ShotBlocker — Apply ShotBlocker
  Arms: ShotBlocker

SUMMARY:
Objective The aim of this study was to evaluate the effects of ShotBlocker administration during measles-mumps-rubella (MMR) vaccination on infants' pain level and mothers' satisfaction.

Method. The study was conducted in a Family Health Center affiliated to the Public Health Directorate of a province in eastern Turkey between August and October 2024 using a randomized controlled experimental design. The study sample consisted of 60 infants who received MMR vaccination (ShotBlocker group: n = 30, control group: n = 30). Infants in the ShotBlocker group received ShotBlocker before vaccine injection, while infants in the control group received only routine vaccine injection. Infant information form, FLACC pain scale and Newcastle Satisfaction with Nursing Care Scale were used for data collection. Ethical principles were followed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* He's 12 months old,
* MMR vaccine will be administered,
* growth-development is normal,
* no analgesic medication was given during the day,
* at least high school graduate
* mothers who volunteered to participate in the study

Exclusion Criteria:

* Neurological disease,
* a chronic disease,
* allergy (egg allergy)
* infants with symptoms of hyperthermia

Ages: 12 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Face, Legs, Activity, Crying, Consolability Pain Scala | pre-test post-test (approximately three months)
  min-max (0-10), lower score means better result, reduce scale scores

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No